CLINICAL TRIAL: NCT02219854
Title: Single-center Study on Laparoscopic Distal Subtotal Gastrectomy for Advanced Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Chief of surgery, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LASS-01
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic gastrectomy (Experimental): Laparoscopic distal subtotal gastrectomy with D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic gastrectomy
- Open gastrectomy (Active Comparator): Open distal subtotal gastrectomy with D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Open gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic gastrectomy
  Arms: Laparoscopic gastrectomy
Procedure: Open gastrectomy
  Arms: Open gastrectomy

SUMMARY:
Laparoscopic distal subtotal gastrectomy with lymph node dissection for treatment of gastric cancer is popular in East Asian countries. However, the long-term follow-up outcome based on randomized clinical trial (RCT) is still rare. Some studies indicated that laparoscopic distal subtotal gastrectomy with D2 lymphadenectomy is a technically feasible and safe procedure by experienced surgeons in high-volume specialized hospitals. However, the application of it is still limited because of lack of solid evidence on the oncologic efficacy. Nowadays, the proportion of patients with locally advanced gastric cancer is estimated up to 80 percent of all gastric cancer cases in China. Before the clinical application of laparoscopic procedure for the treatment with curative intent to advanced gastric cancer located at the middle- or lower-third of the stomach, the oncologic efficacy must be verified.Accordingly, the comparison of long-term outcome between laparoscopic and open distal subtotal gastrectomy with D2 lymphadenectomy for locally advanced gastric cancer based on a well designed RCT is needed.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy cT2-4a, N0-3, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual Seventh Edition Expected curative resection through distal subtotal gastrectomy with D2 lymphadenectomy Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale ASA (American Society of Anesthesiology) score class I, II, or III Written informed consent

Exclusion Criteria:

* Women during pregnancy or breast-feeding Severe mental disorder History of previous upper abdominal surgery (except laparoscopic cholecystectomy) History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging History of other malignant disease within past five years History of previous neoadjuvant chemotherapy or radiotherapy History of unstable angina or myocardial infarction within past six months History of cerebrovascular accident within past six months History of continuous systematic administration of corticosteroids within one month Requirement of simultaneous surgery for other disease Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer FEV1<50% of predicted values

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months

SECONDARY OUTCOMES:
Morbidity | 30 days
3-year overall survival rate | 36 months
3-year recurrence pattern | 36 months
Mortality | 30 days
Morbidity | 36 months
Mortality | 36 months
Postoperative recovery situation | 10 days
  Time to first ambulation, flatus, liquid diet, soft diet and duration of hospital stay are used to assess the postoperative recovery situation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China